CLINICAL TRIAL: NCT02361424
Title: First Single-blind Sequential Placebo-controlled Prospective Phase IIA Pilot Study Assessing the Effects of PXT00864 in Mild AD Patients
Brief Title: Pilot Study Assessing the Effects of PXT00864 in Patients With Mild Alzheimer Disease (AD)
Acronym: PLEODIAL-I
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharnext S.C.A. (Other)
Collaborators: Ascopharm Groupe Novasco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CLN-PXT00864-03
Record Dates: First submitted 2014-12-19; First posted 2015-02-11 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2015-10

CONDITIONS: Alzheimer Disease
Keywords: PXT00864; mild AD; phase 2a
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PXT00864 Dose 1 (Experimental): 1 orange capsule containing 0.4 mg of acamprosate , and 1 white capsule containing 6 mg of baclofen These 2 capsules are taken orally b.i.d. during 8 weeks.
  Interventions: Drug: PXT00864
- PXT00864 Dose 2 (Experimental): 1 orange capsule containing 1 mg of acamprosate , and 1 white capsule containing 15 mg of baclofen .
  These 2 capsules are taken orally b.i.d. during 8 weeks.
  Interventions: Drug: PXT00864
- PXT00864 Dose 3 (Experimental): 1 orange capsule containing 20 mg of acamprosate , and 1 white capsule containing 12 mg of baclofen .
  These 2 capsules are taken orally b.i.d. during 8 weeks.
  Interventions: Drug: PXT00864
- Placebo of PXT00864 (Placebo Comparator): 1 orange capsule containing placebo of acamprosate , and 1 white capsule containing placebo of baclofen .
  These 2 capsules are taken orally b.i.d. during 4 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: PXT00864 — PXT00864 is a fixed-dose combination of baclofen and acamprosate
  Arms: PXT00864 Dose 1; PXT00864 Dose 2; PXT00864 Dose 3
Drug: placebo
  Arms: Placebo of PXT00864

SUMMARY:
The purpose of this study is to assess the safety and efficacy on cognitive impairment and functioning of several doses of PXT00864 (new fixed combination of acamprosate and baclofen at low dose) in patients with mild Alzheimer Disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥ 60 years.
* Patient with a diagnosis of probable AD
* Progressive decline in cognition for more than six months which story is documented in patient medical records
* A Mini-Mental State Examination (MMSE) score of 20-26
* With a minimum of educational background
* Naïve to anti-dementia treatment
* MRI assessment which corroborates the clinical diagnosis (hippocampal atrophy) and excludes other potential causes of dementia especially cerebrovascular lesions
* If available, Cerebral Spinal Fluid (CSF) classical biomarkers should be at levels which corroborate the clinical diagnosis
* Ambulatory patient living at home with a caregiver available and living in the same household or interacting with the patient daily and available if necessary to ensure administration of the investigational product
* Absence of major or severe depressive disease
* Patient with a willingness to participate in this study and who have signed an informed consent form

Exclusion Criteria:

* Early onset of dementia, i.e. before 60 years old to avoid hereditary AD forms
* Significant neurological disease other than AD
* Major psychiatric disorder or syndrome (schizophrenia or bipolar disorder)
* Seizure disorders
* Other infectious, metabolic or systemic diseases affecting central nervous system
* Other active clinically significant illness
* Hospitalization or change of chronic concomitant medications one month prior to screening
* Patients with severe respiratory, hepatic or renal failure or with any other significantly potentially disabling abnormality detected during screening
* Known hypersensitivity to the tested treatment including active substance and excipients.
* Patients participating in another study and exposed to any investigational therapy within the 30 days prior to the entry in this study.
* Patient without medical care insurance

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in the total score of the 11-item Alzheimer´s Disease Assessment Scale- Cognitive Subscale (ADAS-Cog) | Visit V0 (train), V1 (baseline), and every 4 weeks (visits V2, V3 and V4)
  Scores on the ADAS-Cog range from 0-70 with higher scores indicating greater cognitive impairment.
Number of Treatment Emergent Adverse Events (TEAEs) | throughout the 12-week study period.

SECONDARY OUTCOMES:
Change From Baseline in the score of the Digit Symbol Substitution Test (DSST) | Visit V0 (train), V1 (baseline), and every 4 weeks (visits V2, V3 and V4)
  Scores on the DSST range from 0-93 with lower scores indicating greater impairment.
Change From Baseline in the speed to perform the Zazzo's Cancellation Test | Visit V0 (train), V1 (baseline), and every 4 weeks (visits V2, V3 and V4)
Change From Baseline in the score of the Zazzo's Cancellation Test | Visit V0 (train), V1 (baseline), and every 4 weeks (visits V2, V3 and V4)
Change From Baseline in the score of the 15-second Isaacs Set Test | Visit V0 (train), V1 (baseline), and every 4 weeks (visits V2, V3 and V4)
Change From Baseline in the time score of the Trail Making Test - part A | Visit V0 (train), V1 (baseline), and every 4 weeks (visits V2, V3 and V4)
Change From Baseline in the time score of the Trail Making Test - part B | Visit V0 (train), V1 (baseline), and every 4 weeks (visits V2, V3 and V4)
Change From Baseline in the score of the Free and Cued Selective Reminding Test (FCSRT) | 1 (baseline) and V4 (end of study, after 12 weeks of treatment)
  FCSRT is a memory test administered according to the procedure described by Gröber and Buschke modified with 16 verbal items.
Change From Baseline in the score of the 4-item Instrumental Activities of Daily Living scale (IADL-PAQUID) | V0 (train), V1 (baseline), and every 4 weeks (V2, V3 and V4)
  The 4-item Instrumental Activities of Daily Living scale (IADL) concerns four routine daily functions (using transportation, managing finances, using the phone and managing medicines use). Scores on the IADL range from 4-15 with higher scores indicating greater impairment.
Change From Baseline in the score of the Clinical Dementia Rating (CDR) scale | 1 (baseline) and V4 (end of study, after 12 weeks of treatment)
  The Sum of Boxes score of the CDR ranges from 0 to 18, with higher scores indicating greater impairment.
Change From Baseline in the score of the Apathy Inventory (AI) scale | 1 (baseline) and V4 (end of study, after 12 weeks of treatment)
  Scores on the AI range from 0-12 with higher scores indicating greater impairment.

OTHER OUTCOMES:
Change From Baseline in the cognitive Event Related Potential parameters (optional) | V1 (baseline), and every 4 weeks (V2, V3 and V4)
  Some cognitive Event Related Potentials (ERP) with auditory oddball paradigm are performed as an ancillary study.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Orgogozo, MD, Principal Investigator — Hospital Pellegrin, Bordeaux, France
Locations (1):
- CMRR, Bordeaux, France